CLINICAL TRIAL: NCT03970811
Title: Clinical Evaluation of the Effect of Temporization on the Peri-implant Soft Tissue of Immediate Implants: A Randomized Controlled Clinical Trial
Brief Title: Effect of Temporization on the Peri-implant Soft Tissue of Immediate Implants: Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Misr International University (Other)
Collaborators: Zinedent (Unknown)
Responsible Party: Principal Investigator, Shahinaz Elashiry, Associate Professor, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIU-IRB -1819-079
Record Dates: First submitted 2019-05-25; First posted 2019-06-03 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Dental Restoration, Temporary
Keywords: temporization immediate implants peri-implant soft tissue
MeSH Terms: interventions — Dental Restoration, Temporary

STUDY DESIGN:
Intervention Model Description: This parallel arms, randomized controlled clinical trial will involve 22 systemically free patients with an unrestorable tooth in the upper esthetic zone. They will be randomly allocated to two equal groups. Group A (test group) will receive immediate implants with simultaneous immediate temporization, while group B (control group) will receive immediate implants with no temporization.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate implants with immediate temporization (Experimental): Immediate implants with simultaneous immediate placement of temporary crown and placement of the final restoration (loading) will be done 3 months postsurgical
  Interventions: Procedure: Immediate Implants; Procedure: temporary restoration; Procedure: final restoration
- Immediate implants without temporization (Active Comparator): Immediate implants without the use of temporary crown and placement of the final restoration (loading) will be done 3 months postsurgical
  Interventions: Procedure: Immediate Implants; Procedure: final restoration

INTERVENTIONS:
Procedure: Immediate Implants — dental implants are immediately placed after tooth extraction
Procedure: temporary restoration — temporary restoration will be placed immediately after implant placement
  Arms: Immediate implants with immediate temporization
Procedure: final restoration — final restoration (loading) will be placed 3 months postsurgical

SUMMARY:
This parallel arms, randomized controlled clinical trial will involve 22 systemically free patients with an unrestorable tooth in the upper esthetic zone. They will be randomly allocated to two equal groups. Group A (test group) will receive immediate implants with simultaneous immediate temporization, while group B (control group) will receive immediate implants with no temporization. After scaling root planing, the clinical parameters including PES, gingival recession, gingival thickness, postoperative pain and swelling as well as radiographic parameter obtained from Cone Beam Computed Tomography (CBCT) (buccal bone thickness) will be recorded. Immediate implant placement will be performed followed by simultaneous temporization in group A only. Postoperative medication will be prescribed to the patient and postoperative instructions will be explained in detail. Monthly follow-up will be performed to ensure performing proper oral hygiene. Data will be recorded at baseline (at time of implant insertion), three months, six months and nine months post prosthetic placement. Data collected will be tabulated and statistically analysed.

DETAILED DESCRIPTION:
• Intervention:

1. Calibration process: Before beginning the study, outcome assessment will be calibrated. Outcome assessment will be performed by Co-investigator-II and Principal investigator. The calibration process will be repeated until each investigator has substantial correlation as measured by Cohen's Kappa (k ≥ 0.6).
2. Clinical examination and preoperative evaluation using Cone Beam Computed Tomography (CBCT) (Recruitment):

   1. Evaluation of the patient's general condition of the oral cavity, to make sure it complies with the criteria required to be enrolled in the study in terms of oral hygiene, pathological conditions, occlusion and inter-arch space.
   2. Evaluation of the soft tissue biotype by trans-gingival piercing using a periodontal probe.
   3. Width of keratinized gingiva in millimeters (measured by a periodontal probe from the gingival margin to the mucogingival junction). It is measured at three areas (mesial, mid buccal and distal)
   4. A preoperative CBCT will be performed for all patients before enrollment as a standard procedure. Evaluation and recording of the periapical condition, crestal bone level, available buccal bone thickness (not less than one millimeter), bucco-palatal bone width, height and density. Suitable implant length and diameter will be determined as well.

   Patients with all inclusion criteria will be offered to participate in the study and sign a consent form.
3. Random allocation: After consenting, each patient will be allocated in one of the two study groups randomly using random numbers generated by rand.org created and kept by a teaching assistant not participating in the study. Grouping will be as follows:

   * Group A (test group): Immediate implants placed with simultaneous immediate temporization (Immediate Implants + Immediate Temporization).
   * Group B (control group): Immediate implants only
4. Allocation concealment: It will achieved using a sealed coded opaque envelopes containing treatment of the subject. They will be kept by the teaching assistant. The envelope will be handed to the principal investigator and opened just before performing the surgical procedure.
5. Blinding: blinding of investigators, outcome assessors and participants cannot be achieved due to the presence of a temporary crown in test group immediately after implant placement while being absent in the control group.
6. Surgical procedure:

   Surgical procedures will be carried out by Co-invesigator-I. Following the administration of local anesthesia, atraumatic extraction will be done using a remaining root or anterior forceps.

   After proper curettage of the socket wall using a small bone curette to remove any granulation tissue, implant insertion is performed according to manufacturer's instructions as follows:
   * A point of entrance for the drills will be created using a surgical round bur.
   * Drills will be used sequentially until the required implant diameter is reached.
   * Implant insertion will be done in the osteotomy site using a torque wrench by self-tapping fashion till the implant is leveled about two mm apical to the alveolar bone crest with adequate primary stability (torque above 35N).
   * After implant placement, a periapical radiograph using a radiographic holder and a radiographic stent will be taken to determine the crestal bone level. The parallel technique in combination with the acrylic stent will be used to ensure reproducibility.

   As regards the control Group (Group B), no temporization is needed. Implant exposure and subsequent prosthetic placement of the final restoration (loading) will be performed 3 months postsurgical. As for the test group (Gp A), temporization procedures will be done immediately after implant placement utilizing a temporary abutment supplied by the manufacturer which will be scanned once placed using an intraoral scanner [Dentsply blue cam]. Designing will be performed using Inlab premium 4.4 software. Milling of the provisional crowns will done using CEREC [Dentsply] with estimated milling time of 25 minutes per crown. Polymethylmethaacrylate (PMMA) blanks will be used to fabricate the provisional crowns. Crowns will be finished and polished by Soflex finishing and polishing kits. Adequate emergence profile, marginal fit, occlusion and esthetics will be confirmed and the occlusion will refined using medium then fine articulating paper. Final repolishing is mandatory to ensure absence of gingival inflammation.
7. Postoperative Care:

   1. Antibiotics (Amoxicillin 1g orally- twice daily for 5 days).
   2. Anti-inflammatory drugs (NSAIDS; Ibuprofen 600mg three times daily after meals for 5 days).
   3. Antiseptic mouthwash (0.12% Chlorhexidine) will be prescribed for 60 seconds, 15 ml each time, two times a day for 14 days.
   4. Patient self-care instructions:

      * Application of an ice bag to the treated area for the first 24 hours.
      * Gently brushing the operated area starting from the second day with a soft brush using roll technique.
8. Follow-up: Patients' recall visits will be scheduled every month for supportive periodontal therapy and recording of outcome variables at three, six and nine months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have at least one unrestorable tooth in the upper esthetic zone (anterior teeth and premolars) that need to be extracted with sound neighboring teeth
2. Systemically free patients (American Society of Anesthesiologists I)
3. Patients aged from 18 to 65 years old
4. Buccal bone thickness should be at least 1mm assessed in CBCT
5. Sinus floor or nasal floor clearance from root apex at least 4 mm as assessed in CBCT
6. Good oral hygiene
7. Accepts nine months follow-up period (cooperative patients)
8. Patient accepts to provides an informed consent

Exclusion Criteria:

1. Patients with signs of acute infection related to the area of interest or any pathological lesions that affect healing
2. Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits such as bruxism
3. Smokers
4. Pregnant and lactating females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-22 (Estimated)

PRIMARY OUTCOMES:
change in Pink Esthetic Score (PES) | at 3, 6, 9 months
  This will be performed by outcome assessor. PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score. The mesial and distal papilla will be evaluated for completeness, incompleteness or absence. All other variables will be assessed by comparison to a reference tooth (contralateral tooth).

SECONDARY OUTCOMES:
White Esthetic Score (WES) | at 9 months
  This will be performed by outcome assessor. WES focuses on the visible part of the implant restoration based on five parameters: general tooth form, outline, clinical crown volume, color including (hue and value), surface texture, translucency and characterization. a score of 2,1,0 is assigned to the five parameters. All the five parameters will be assessed by direct comparison with the contralateral reference tooth.

OTHER OUTCOMES:
change in Gingival recession | at 3, 6, 9 months
  This will be performed by outcome assessor by measuring distance from gingival margin to the implant platform in mm using University of North Carolina (UNC)15 periodontal probe.
change in Gingival thickness | at 3, 6, 9 months
  This will be performed by outcome assessor by piercing gingival tissues horizontally, perpendicular to the long axis of the tooth/implant until it contacts bone, at 9 different points; three readings: mesially, mid buccally and distally at three different levels; 2mm, 4mm and 6mm apical to the gingival margin. The length of the part of the instrument that penetrated into the soft tissue is measured in mm. This will be done using anesthetic needle with a rubber stopper added.
change in Post-operative pain | daily for 14 days, starting day of surgery
  Recorded by the patient using a Visual analogue scale (VAS) scale, where (1) indicates the least pain and (10) indicates the worse pain. It will be done by the patient starting day of surgery and for 14 days (always taken before bedtime at a fixed time point for each patient).
change in Post-operative swelling | daily for 7 days, starting day of surgery
  Recorded by the patient using using a Visual analogue scale (VAS) scale, where (1) indicates the mild swelling and (10) indicates the severe swelling. It will be always taken before bedtime at a fixed time point for each patient.
  Numerical values will be transformed to categories by outcome assessor as follows:
  0= absent (no swelling) 1-3= slight intraoral swelling at the operational area 4-6= moderate intraoral swelling at the operational area 7-10= intense extraoral swelling extending beyond the operational area
change in Buccal bone thickness at different levels | presurgical (for inclusion in the study), at 9 months
  This will be performed by outcome assessor mid bucal at 0, 2, 4 and 6 mm from the crest of bone presurgical and at 9 months.
Patient satisfaction | at 9 months
  Performed by the patient filling a 3-item questionnaire where the patients is asked to use a 5 point answer scale.

CONTACTS AND LOCATIONS:
Overall Officials: Shahinaz G Elashiry, Assoc. Prof., Principal Investigator — Periodontics Dep., Faculty of Dentistry, Misr International University; Hani El-Nahass, Assoc. Prof., Study Director — Periodontics Dep., Faculty of Dentistry, Cairo University; Fatma H Eldemerdash, Lecturer, Study Chair — Periodontics Dep., Faculty of Dentistry, Misr International University; Talaat Samhan, Lecturer, Study Chair — Fixed Prosthodontic Div., Faculty of Dentistry, Misr International University
Locations (1):
- Misr International university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No